CLINICAL TRIAL: NCT05218044
Title: Cryoablation as a Minimally Invasive Alternative to Surgery for Managing Ductal Carcinoma In Situ
Acronym: DCIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glendale Adventist Medical Center d/b/a Adventist Health Glendale (Other)
Collaborators: Helen Rey Breast Cancer Research Foundation (Unknown); California Oncology Research Institute (Unknown); Doterra Healing Hands Foundation (Unknown)
Responsible Party: Principal Investigator, Dennis Holmes, Principal Investigator, Glendale Adventist Medical Center d/b/a Adventist Health Glendale
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIS Cryo
Record Dates: First submitted 2021-12-23; First posted 2022-02-01 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Ductal Carcinoma in Situ
Keywords: DCIS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Cryosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryoablation (Other): Phase I, single-arm study to evaluate the ability of cryoablation to achieve complete ablation of DCIS in the cryoablation zone of necrosis as a potential alternative to surgery.
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — The cryoprobe tip will be inserted into the breast and directed under ultrasound guidance to the location where the ultrasound visible marker is located. Next, the cryoprobe will be used to freeze a 4 X 3 X 3 cm diameter area of DCIS using two separate 10-minute freeze cycles separated by a single 10-minute thaw cycle. The cryoprobe will remain in place the entire time. After the second freeze, the cryoprobe will be withdrawn from the breast and a bandage will be applied to the skin.

SUMMARY:
Cryoablation or tumor freezing is a percutaneous, office-based procedure that is emerging as a minimally invasive, cost-effective alternative to surgery that is currently being evaluated in clinical trials for the management of for early-stage invasive breast cancer. The investigator will also evaluate the potential of cryoablation as a minimally invasive alternative to surgery for small areas of DCIS by examining its ability to achieve complete ablation of DCIS within the targeted cryoablation zone of necrosis.

ELIGIBILITY:
Inclusion Criteria:

* DCIS spanning 2 cm or less based on its radiographic appearance by mammography and/or breast contrast-enhanced MRI
* Diagnosis of DCIS by minimally invasive needle biopsy
* No prior history of DCIS or invasive breast cancer in the same breast
* No history of surgical biopsy and/or lumpectomy for diagnosis/treatment in the same breast
* Adequate breast volume and skin clearance to permit cryoablation as assessed by Dr. Holmes. This excludes male and females with breasts too small to allow safe cryoablation
* Non-pregnant, non-lactating, and no history of pregnancy within the preceding 6 months
* No history of breast radiation in the same breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Ability of cryoablation to achieve complete ablation of DCIS | 6 months
  Number of participants to achieve completeness of ablation by measuring the percentage of subjects with no residual DCIS or invasive cancer within the zero of necrosis assessed in the post-cryoablation core biopsy obtained 6 months post-cryoablation.

SECONDARY OUTCOMES:
Recurrence rate | 5 years
  Number of participants at the 5-year rate of invasive breast cancer recurrence after cryoablation of DCIS measuring </= 2cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Office of Dennis R. Holmes, M.D., F.A.C.S., Glendale, California, United States